CLINICAL TRIAL: NCT02010580
Title: The Effects of Vaginal Ospemifene on Pelvic Organ Vascularity and Blood Flow in Postmenopausal Women
Brief Title: Effects of Ospemifene on Pelvic Vascularity and Blood Flow
Acronym: Osphena
Status: Withdrawn | Type: Observational
Why Stopped: Never received necessary funding.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 3555
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osphena: Subjects will be randomized in a ratio of 1:1 to receive either 60 mg of ospemifene (Osphena, Shionogi, Florham, NJ) or placebo tablet.

SUMMARY:
Subjects will be randomized in a ratio of 1:1 to receive either 60 mg of ospemifene (Osphena, Shionogi, Florham, NJ) or placebo tablet. Placebo tablets will be identical in appearance and packaging will be identical for the two pills. The participants will be instructed to take one tablet in the morning with food for twelve weeks. Basic demographic information will be obtained on all participants. All women will undergo a pelvic examination, and questionnaires regarding pelvic floor dysfunction and sexual function before and three months after treatment. 3-D ultrasound with Doppler blood flow analysis will be performed before the patient is started on the treatment. 3 months after treatment, the 3-D ultrasound with Doppler blood flow analysis will be repeated. Four areas will be measured:

1. The urethra in exactly the same section at the same level with the same setups.
2. 3 and 9 O'clock position
3. 6 o'clock position
4. Clitoral blood flow Doppler blood flow will be visualized using the Doppler color mode of the ultrasound machine and will be applied for the assessment of the vascularity pattern. Additionally, we will record a film with the use of Color Doppler in a video file. The transducer will be immobilized at one selected section and record a ten seconds of film. This film will be further analyzed in special software called Pixel flux after the examination. Dr. Pawel Wieczorek and Dr. Magdalena Wozniak will read these deidentified video files in a randomized fashion based on their previous research experience with similar video interpretations of pelvic color Doppler imaging [8-11].

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Available for reliable follow up
* Able to complete study assessment
* Mammogram within the last year
* Menopausal (at least 12 months since last spontaneous menstrual bleeding)

Exclusion Criteria:

* Age <18 years
* Dementia or inability to follow instructions
* Prior pelvic floor radiation
* History of uterine, ovarian, fallopian tube, breast, or colon cancer
* Current use or use within the last 6 months of estrogen (vaginal, oral, transdermal, compounded)
* Current use of alternative medicines including black cohosh, evening primrose, dong quai, or chasteberry
* Known prothrombotic mutations such as Factor V Leiden, prothrombin mutation, protein C or Protein S deficiency
* History of or current thrombophelbitis or venous thromboembolic disorders
* Currently using fluconazole or rifampin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We estimate that we will need a total of 30 patients recruited to this study. Eligible subjects will be postmenopausal women who have undergone menopause and have had a hysterectomy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Doppler Flow Analysis | 3 months post-treatment
  To prospectively evaluate, by three-dimensional (3-D) Doppler flow analysis, the hemodynamic vaginal blood flow variations between women receiving oral ospemifene versus women receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Shobeiri, MD, Principal Investigator — University of Oklahoma